CLINICAL TRIAL: NCT06580119
Title: Potential Benefits of the Somatic Psychoeducational Intervention for Improving Health and Wellness
Brief Title: Somatic Psychoeducational Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB202401217
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Work Related Stress
Keywords: Polyvagal Theory; Stress; Trauma; Neuroendocrine Biomarkers; Somatic Intervention; Oxytocin; PTSD; Mental Health; Neuroendocrine Functioning; Physical Health; Emotional Health; Coping Behaviors; Mindfulness; Burnout; Tai Chi; Psychoeducation; Breathing Exercises
MeSH Terms: conditions — Occupational Stress; Wounds and Injuries; Stress Disorders, Post-Traumatic; Psychological Well-Being; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: The participants will be assigned to Group A or Group B. Intervention Group A will be provided the in-person intervention and Group B will be provided the virtual.
  During Phase 1, Group A will receive the intervention and Group B will act as the control group. During Phase 2, Group B will receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: In-Person (Experimental): Participants will be asked to participate in the 4 intervention classes in person. The pre-intervention and post-intervention assessments will require participants to complete a 20-25-minute online survey via Qualtrics and provide saliva samples.
  Interventions: Behavioral: Somatic Psychoeducational Intervention
- Group B: Virtual (Active Comparator): Participants will be asked to participate in the 4 intervention classes virtually. The pre-intervention and post-intervention assessments will require participants to complete a 20-25-minute online survey via Qualtrics and provide saliva samples.
  Interventions: Behavioral: Somatic Psychoeducational Intervention

INTERVENTIONS:
Behavioral: Somatic Psychoeducational Intervention — Participants will work on increasing bodily awareness by learning psychoeducation, movement techniques, and relaxation.

SUMMARY:
The goal of this clinical trial is to explore possible benefits and mechanisms through which the Somatic Psychoeducational Intervention can improve health and wellness. The main goals of the study are:

* To understand how the participants are doing with regard to their mindfulness, coping behaviors, emotional, physical, and work health, and autonomic reactivity (the degree participants physiologically respond).
* To examine regulation of the oxytocinergic system
* To investigate whether pre-intervention measures relate to the overall functioning
* To determine the 1-week and 1-month post-intervention effects of the Intervention(s)
* To identify individual characteristics that influence the effectiveness of the intervention at the 1-week and 1-month post-intervention assessments.

Participants will:

* complete the online pre-assessment measures regarding how they are doing emotionally and with respect to their work situation.
* listen to 15-minutes of calming music and provide pre and post-music salivary samples
* complete pre-intervention, post-intervention, 1-week post-intervention, and 1-month post-intervention assessments that involve completion of online measures and collection of saliva samples.
* participate in the intervention (which involves 4 hours; the 1-hour classes will be administered over four weeks).

Researchers will compare the Intervention Group A (in-person) to Intervention Group B (virtual) to see if the Intervention Group A experiences greater improvements in their health and wellness.

DETAILED DESCRIPTION:
It is the intent of this proposal to experimentally explore the possible benefits and mechanisms through which the Somatic Psychoeducational Intervention can influence emotional and physical health and autonomic and neuroendocrine functioning. This will be accomplished by our team by using well-validated self-report measures of mental health and autonomic reactivity and non-invasive measurements of levels of oxytocin.

Specific Aims:

* Specific Aim 1: To investigate whether participants who have difficulty regulation of the oxytocinergic system after listening to calming music relate to the overall functioning of the participants.
* Specific Aim 2: To investigate whether pre-intervention measures of autonomic reactivity and the neuropeptides oxytocin relate to the overall functioning of the participants
* Specific Aim 3: To determine if the intervention leads to improvements in functioning post, 1-week post, and 1-month post the Intervention
* Specific Aim 4: To identify individual characteristics that influence the effectiveness of the intervention post, 1-week post, and 1-month post intervention.

Experimental design

* The participants will be randomly assigned to either Group A or Group B. Intervention Group A will be provided the intervention in-person. Group B will be provided the intervention virtually.
* The invited participants will listen to 15-minutes of calming music via headphones pre-intervention to examine the regulation of the oxytocinergic system via providing pre and post music salivary samples. The participants will be provided the option to wear an eye mask while listening to the music to help them focus on the music.
* The invited participants will complete assessments immediately before the intervention, immediately after the intervention, 1 week after the intervention, and 1 month after the intervention. Assessments involve online measure and collection of saliva samples.
* The Somatic Psychoeducational Intervention will be provided in four classes, and the participants will be awarded for their time financially.
* Between-subject analyses will compare the session 1 data to determine if the participants in Group A exhibit greater improvements than the participants in Intervention Group B. Within-subject repeated measures analyses will determine the potential benefits of the intervention for all participants by comparing their functioning at the various time points.

  * For the outcome measures, change scores will be calculated to determine the change from the pre-intervention to the post intervention assessment, change from the pre-intervention to the 1-week post-intervention assessment, and from the 1-week post-intervention assessment to the 1-month post-intervention assessment. These changes scores will be used to determine if there are pre-intervention factors that impact the success of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Individuals are eligible to participate if they are between 18 and 89 years old and are providers at the Jewish Family & Community Services (JFCS)

Exclusion Criteria:

* Individuals are not eligible to participate if they are under 18 years old or older than 89 years old

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Measuring Change in Depressive Symptoms using the Patient Health Questionnaire (PHQ-8) self-report questionnaire. | Baseline up to 1-month (post-intervention)
  Depression
Measuring Change in anxiety using the General Anxiety Disorder 7 self-report questionnaire. | Baseline up to 1-month (post-intervention)
  Anxiety
Measuring Change in autonomic reactivity using the Body Perception Questionnaire self-report questionnaire. | Baseline up to 1-month (post-intervention)
  Autonomic Reactivity
Measuring Change in social engagement using the Neuroception of Psychological Safety Scale self-report questionnaire. | Baseline up to 1-month (post-intervention)
  Social Engagement
Measuring Change in Posttraumatic Stress Symptoms using the Posttraumatic Stress Disorder Checklist 5 self-report questionnaire. | Baseline up to 1-month (post-intervention)
  Posttraumatic Stress Symptoms
Measuring Change in Mindfulness using the Five Facets of Mindfulness self-report questionnaire. | Baseline up to 1-month (post-intervention)
  Mindfulness
Measuring impact of prior adversity using the Adverse and Traumatic Experiences Scale self-report questionnaire. | Baseline up to 1-month (post-intervention)
  Prior Adversity
Measuring change of professional health outcomes using self-report questionnaires. | Baseline up to 1-month (post-intervention)
  Professional Fulfillment, burnout, and retention
Measuring change in neuroendocrine functioning | Baseline up to 1-month (post-intervention)
  Oxytocin Levels

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes P Dale, PhD, Principal Investigator — University of Florida
Locations (1):
- The LJD Jewish Family & Community Services (JFCS) Headquarters, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dale LP, Dana AN, Lamont H, Nazarloo P, Carter CS, Porges SW, Cuffe SP, Van Vleet Goelz D. Somatic Psychoeducational Intervention Is Associated with Increased Oxytocin Levels, Improved Autonomic Function, and Reduced Psychological Distress Symptoms in Medical and Social Care Professionals. Healthcare (Basel). 2025 Dec 10;13(24):3236. doi: 10.3390/healthcare13243236. PMID 41464305